CLINICAL TRIAL: NCT03023748
Title: Providing Intravenous Paricalcitol Treatment to the Sick and Poor Chronic Hemodialysis Patients With Severe Secondary Hyperparathyroidism Resistant to Existing Vitamin D Analogs
Brief Title: Intravenous Paricalcitol in Chronic Hemodialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Dr. Angela Yee-Moon Wang, Honorary Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW11-293
Record Dates: First submitted 2017-01-07; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Endstage Renal Disease; Secondary Hyperparathyroidism
Keywords: activated vitamin D treatment
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intravenous paricalcitol solutions (Experimental): Intravenous paricalcitol will be administered twice or thrice weekly post-hemodialysis with a dose based on the baseline iPTH level divided by 120.
  For instance, with a baseline iPTH 1200pg/mL, an induction dose of 10mcg twice or thrice weekly will be given. The maximum weekly dose allowed is 30mcg. Subsequent dose titration may be required depending on the serum PTH level. Intravenous paricalcitol will be continued up to 24 months.
  Interventions: Drug: Intravenous Paricalcitol

INTERVENTIONS:
Drug: Intravenous Paricalcitol — Twenty four months of intravenous paricalcitol will be given twice or thrice weekly post-hemodialysis depending on frequency of hemodialysis of the patients
  Other Names: Zemplar

SUMMARY:
This study aims to provide intravenous paritcalcitol treatment for the sick and poor hemodialysis patients with severe secondary hyperparathyroidism (SHPT) resistant to existing vitamin D analogs therapy or with hypercalcemia precluding the use of existing vitamin D analogs.

The study aims to evaluate the effect of paricalcitol on control of SHPT, biochemical parameters of chronic kidney disease-mineral bone disease, cardiac parameters, vascular calcification and stiffness parameters and nutrition status in patients receiving chronic hemodialysis treatment.

DETAILED DESCRIPTION:
This is a 2-year single-arm intervention study of which intravenous paricalcitol will be provided as a second-line treatment to 30 chronic hemodialysis patients with severe SHPT (defined as intact parathyroid hormone [iPTH] ≥ 800pg/mL) resistant to existing vitamin D analogs treatment (including rocaltrol and alfacalcidol) or with hypercalcemia (defined as serum calcium ≥2.56mmol/L) precluding the use of existing vitamin D analogs.

The study aims to evaluate the control of SHPT, various biochemical parameters of chronic kidney disease-mineral bone disease, left ventricular mass and volumes, vascular calcification and stiffness parameters, handgrip strength and serum albumin with the use of intravenous paricalcitol in patients receiving chronic hemodialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients with severe SHPT (defined as iPTH ≥ 800pg/mL) resistant to rocaltrol or alfacalcidol (defined as iPTH not controlled in the range between 2 - 9 times of lab upper limit reference).
* Chronic hemodialysis patients with severe SHPT and at the same time hypercalcemia (defined as serum calcium ≥2.56mmol/L) but still < 2.8mmol/L precluding the use of rocaltrol or alfacalcidol but still feasible to use paricalcitol.

Exclusion Criteria:

* Patients with metastatic malignancy,
* Patients with extremely poor general condition (eg. bedbound) and expected lifespan is below 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular mass index | 52 weeks and 104 weeks
  MRI determined cardiac parameters

SECONDARY OUTCOMES:
Change in Coronary artery calcium score | 52 and 104 weeks
  Computed tomography determined coronary artery calcium score
Change in Aortic stiffness | 52 and 104 weeks
  aortic pulse wave velocity
Change in handgrip strength | 52 and 104 weeks
  nutrition and functional parameters
Change in Serum albumin | 52 and 104 weeks
  Nutrition parameters
Change in serum Calcium and phosphate | 52 and 104 weeks
  Biochemical parameters of CKD-MBD
Change in Intact parathyroid hormone | 52 and 104 weeks
  Biochemical parameters of CKD-MBD
Change in alkaline phosphatase | 52 and 104 weeks
  biochemical parameters of CKD-MBD

CONTACTS AND LOCATIONS:
Overall Officials: Angela YM Wang, MD PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital and Tung Wah Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No